CLINICAL TRIAL: NCT07154719
Title: GLP-1R Actions on Muscle and the Skeleton
Acronym: GRAMS
Status: Not yet recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Pennington Biomedical Research Center (Other)
Responsible Party: Principal Investigator, Robert Dubin, Principle Investigator, Pennington Biomedical Research Center
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: PBRC 2024-031
Record Dates: First submitted 2025-08-22; First posted 2025-09-04 (Actual); Last update posted 2025-09-04 (Actual); Status verified 2025-08

CONDITIONS: Musculoskeletal Abnormalities; Obesity; Sarcopenic Obesity; Osteoporosis; Drug Effect
Keywords: GLP-1 agonists; Obesity treatments; Muscleskeletal loss; Tirzepatide
MeSH Terms: conditions — Musculoskeletal Abnormalities; Obesity; Osteoporosis | interventions — Tirzepatide

STUDY DESIGN:
Intervention Model Description: The investigators will enroll 25 subjects in each study arm. Both arms will involve treatment with a GLP-1 agonist (tirzepatide) for 5 months.
  The intervention arm will use a lifestyle toolkit which includes protein supplements and resistance-based exercises.
  The control group will use regular diet and exercise activities. Testing includes DXA and MRI body composition as well as lab tests to assess for muscle skeletal quality and physical fitness.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- Treatment/intervention group (Experimental): Treatment with Tirzepatide for 5 months and lifestyle toolkit.
  Interventions: Drug: Tirzepatide
- Control/Placebo (Placebo Comparator): Treatment with Tirzepatide for 5 months with regular diet and exercise.
  Interventions: Behavioral: Lifestyle toolkit

INTERVENTIONS:
Drug: Tirzepatide — GLP-1 based treatment for obesity
  Arms: Treatment/intervention group
Behavioral: Lifestyle toolkit — 2 ABBOTT protein shakes daily and resistance-based exercise x 3 days per week.
  Arms: Control/Placebo

SUMMARY:
The GRAMS study objectives are to assess the musculoskeletal changes that occur after weight loss using GLP-1 based therapy. A lifestyle intervention with diet and exercise is included to assess any mitigating effects are provided, versus a control group with regular exercise and diet.

DETAILED DESCRIPTION:
Obesity and type 2 diabetes remain at epidemic proportions in our country particularly in vulnerable populations such as elderly, and minority patients. Over the last 20 years, the use of incretin-based agents (Glucagon-like Peptide 1 Receptor Agonist (GLP-1 RA) and Glucose dependent insulinotrophic polypeptide (GIP) to treat these disorders has offered unprecedented advances based on significant weight loss and reduction in major cardiovascular endpoints. Whilst weight loss provides a vital aspect for addressing obesity and type 2 diabetes, there are concerns associated with the quality of weight reduction.

The impact of losing weight on the musculoskeletal system has garnered recent attention in the lay press. Reported high-impact studies have reported excessive loss of skeletal muscle using GLP-1 RAs. The data regarding combined therapies (GLP-1 RA and GIP) suggested smaller loses. This preliminary data is based on using a surrogate marker (fat-free mass) determined by dual energy x-ray absorptiometry (DXA).

Recent reviews evaluating the impact that incretin-based agents have on fat-free-mass were found to be inconclusive based on high variability and multiple confounding factors. Assessing the impact that these agents have on the musculoskeletal system is now an important endeavor. (Aim 1-2) Diet-induced weight loss is also associated with bone loss, although little attention has focused on this potentially problematic outcome. In the CALERIE study, modest caloric restriction (15%) over two years led to weight loss and a 2% reduction in hip bone mineral density (BMD) among normal weight individuals. The mechanisms of weight loss-induced bone loss are unclear, although a drop in fat-free mass (which is composed of skeletal muscle, organs, water and connective tissues) principally muscle, such as occurs with the GLP1RAs, may predispose to injury, disability and bone loss. Another possibility is a mechanical form of skeletal adaptation to lower lean mass, through myokine mediated bone remodeling. However, significant trabecular bone loss in a non-weight bearing skeletal site occurs in mice as the investigators have shown in the mandible, from a 30% CR diet (Liu, personal communication). As such gravitational unloading due to weight loss is not solely responsible for deleterious skeletal changes. Despite the dramatic weight and lean mass loss from the GLP1 RAs, few clinical trials have focused on loss of muscle mass and fewer on any skeletal changes. In those that did, the results suggest equipoise for skeletal changes. There are no data on the skeletal effects from tirzepatide which can drive up to 25% weight loss. (Aim 1c) Also, it is unknown whether the addition of dietary modifications and resistance-based exercises impacts skeletal adaptation, muscle mass and bone loss. (Aim 2) Furthermore, there are inconsistent data in non-Hispanic Blacks with the GLP1 RAs because trial participation in under-represented populations has been poor. Hence, there is a major knowledge gap in our understanding the impact that a mixed GIP and GLP1RA, tirzepatide affects muscle and bone mass, particularly among underserved populations.

The wide-spread usage of GLP-1 related agents has not required formal recommendations regarding the use of exercises, specifically resistance-based exercises, or dietary protein optimization to address the potential for loss of fat-free mass or bone mineral density that has been suggested in studies evaluating body composition and bone density in subjects using these compounds. While the data for using such lifestyle interventions with diet and bariatric surgery have confirmed benefits in reducing loss of fat-free mass, the investigators know of only 1 published report using GLP-1 agents and exercise: Lundgren et al. found that in subjects using additional resistance-based exercise had a more favorable impact on sparing fat-free mass.

Additional gaps in our understanding remain despite the growing use and popularity of these agents. Additionally, patients with obesity and type 2 diabetes tend to develop ectopic fat within muscle (myosteatosis) that is not measured as part of fat free mass by DXA. It is posited that the major depot for acute loss of skeletal muscle from rapid weight loss may be from this portion of poor-quality lipid-rich tissue quelling major concerns. (Aim 2b) Aim 3, an explorative outcome, the investigators will determine if tirzepatide causes bone loss by measuring bone formation (P1NP) and bone resorption markers (NTx), if imbalanced skeletal remodeling is related to the change in total lean mass, muscle mass through reduced myokine (i.e., irisin) release, skeletal adaptation to weight change or another endocrine mechanism. Using a team science approach, the investigators will combine the expertise in metabolism and body composition of the PBRC group with skeletal expertise from MaineHealth to provide key insights into musculoskeletal effects from tirzepatide, a relatively new but often sought after drug for weight loss and type 2 diabetes. This supplement could also shed light on newer mechanisms of weight loss-induced bone loss and set the stage for a larger clinical trial.

ELIGIBILITY:
Inclusion Criteria:

* Subjects will have a BMI between 30kg/m2

  * 40kg/m2 (inclusive)
* Be between 18 and 50 years of age (inclusive).
* Non-Hispanic Black males and females will be enrolled at PBRC.
* Rural males and females will be enrolled at MaineHealth.
* Female subjects will be premenopausal.
* Females have had their last menstrual period less than 60 days before screening.
* Females have the absence of menopausal-associated vasomotor symptoms.
* All subjects must be able to use Lifestyle Toolkit as prescribed for intervention arm.

Exclusion Criteria:

- Males and females over the age of 50 years of age

* Menopausal females.
* Subjects on systemic corticosteroids or other agents known to increase loss of muscle and bone mass.
* Subjects who are on medications that increase or decrease weight status.
* Subjects having contraindications to tirzepatide in the package insert.
* Subjects with a history of malignancy other than non-melanoma skin cancer
* Subjects with known osteoporosis or are on osteoporosis therapies (gonadal hormones or hormone antagonists).
* Subjects with uncontrolled thyroid or parathyroid disease that may influence the study results.
* Subjects with a clinically significant hematologic abnormality, kidney disease, liver disease, or diabetes.
* Females of childbearing potential who do not agree to using an effective method of contraception during the study. Medically acceptable methods include oral contraceptive medication, an intrauterine device (IUD), an implantable contraceptive (such as Implanon), or a barrier method (such as condom or diaphragm with spermicide).

Injectable contraceptives such as Depo-Provera are a cause for exclusion in that they can cause bone loss.

Abstinence is acceptable, as is sexual activity exclusively with same sex partners.

Fertility Appreciation Based Methods (natural family planning) are also acceptable forms of addressing childbearing potential in all subjects. A urine pregnancy test (UPT) will be performed on all females of childbearing potential at the screening visit, 3 and 6 months.

* Unable to follow Lifestyle Toolkit as prescribed for intervention arm.
* Patient Health Questionnaire-9 (PHQ-9) Score equal to or greater than 15 (clinical depression).
* Adults who are unable to consent.
* Individuals who are not yet adults (infants, children and teenagers).
* Pregnant females.
* Incarcerated individuals.
* Contraindication to MRI - including but not limited to non-removable metallic or electronic implants, claustrophobia or other fear of confinement, inability to tolerate loud scanner noise, body weight greater than 500 pounds.
* Subjects with a baseline level of 25-OH vitamin D <15 ng/ml will be excluded from the trial. The subject's physician will be notified, and the subject will be referred to their primary care physician.
* Any significant EKG abnormalities that are considered a risk for utilizing weight management therapies.

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 50 (Estimated)
Dates: Start 2025-09-01 (Estimated); Primary Completion 2026-03-01 (Estimated); Study Completion 2026-04-01 (Estimated)

PRIMARY OUTCOMES:
Changes in fat free mass (FFM) using DXA imaging. FFM equals all body composition that is not fat mass. This includes bone, skeletal muscle, organs, water and all connective tissues. The unit of measurement is in kilograms (kg) at baseline, 3 and 6 mo. | Baseline and time 3, and 6 months.
  DXA (Dual energy Xray absorptiometry)

SECONDARY OUTCOMES:
MRI (thigh) without contrast | At baseline, 3 and 6 months
  To assess for muscle quality (% of skeletal muscle to intermuscular fat)
lab tests | baseline and 5 months
  bone markers, micronutrient panel.

CONTACTS AND LOCATIONS:
Locations (1):
- Robert L. Dubin, MD, Baton Rouge, Louisiana, United States

IPD SHARING:
Plan to Share IPD: Yes
Sharing plan of data will be completed by primary study team by 12/01/25. All details will be provided by PI and study team.
Supporting Information: Study Protocol, SAP, ICF, CSR
Time Frame: Data available 2-3 months after study completion date.
Access Criteria: Requests for data sharing can be made to study PI (Dubin). The investigators will provide available data using the available resources at the study center.
URL: http://pbrc.com

REFERENCES:
- [Background] Goodpaster BH, Theriault R, Watkins SC, Kelley DE. Intramuscular lipid content is increased in obesity and decreased by weight loss. Metabolism. 2000 Apr;49(4):467-72. doi: 10.1016/s0026-0495(00)80010-4. PMID 10778870
- [Background] Lundgren JR, Janus C, Jensen SBK, Juhl CR, Olsen LM, Christensen RM, Svane MS, Bandholm T, Bojsen-Moller KN, Blond MB, Jensen JB, Stallknecht BM, Holst JJ, Madsbad S, Torekov SS. Healthy Weight Loss Maintenance with Exercise, Liraglutide, or Both Combined. N Engl J Med. 2021 May 6;384(18):1719-1730. doi: 10.1056/NEJMoa2028198. PMID 33951361
- [Background] Jastreboff AM, Aronne LJ, Ahmad NN, Wharton S, Connery L, Alves B, Kiyosue A, Zhang S, Liu B, Bunck MC, Stefanski A; SURMOUNT-1 Investigators. Tirzepatide Once Weekly for the Treatment of Obesity. N Engl J Med. 2022 Jul 21;387(3):205-216. doi: 10.1056/NEJMoa2206038. Epub 2022 Jun 4. PMID 35658024
- [Background] Dubin RL, Heymsfield SB, Ravussin E, Greenway FL. Glucagon-like peptide-1 receptor agonist-based agents and weight loss composition: Filling the gaps. Diabetes Obes Metab. 2024 Dec;26(12):5503-5518. doi: 10.1111/dom.15913. Epub 2024 Sep 30. PMID 39344838